CLINICAL TRIAL: NCT01185405
Title: Prediction and Adjustment of Voriconazole Plasma Level in Critically Ill Patients
Brief Title: Voriconazole Plasma Level in Intensive Care Unit (ICU) Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sang-Ho Choi, Doctor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVORI
Record Dates: First submitted 2010-08-17; First posted 2010-08-20 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Invasive Fungal Infection
Keywords: Voriconazole; Therapeutic drug monitoring; Intensive care unit
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EA group (Experimental): Voriconazole dosage adjustment according to the each measurements of voriconazole levels from day 1, using NONMEM program
  Interventions: Other: Use of different strategy for voriconazole dosage adjustment
- CA group (Active Comparator): Voriconazole dosage adjustment according to the levels from day 5, using predefined protocol
  Interventions: Other: Use of different strategy for voriconazole dosage adjustment

INTERVENTIONS:
Other: Use of different strategy for voriconazole dosage adjustment — Patients will be randomly assigned into 2 groups: conventional adjustment group (CA group) and early adjustment group (EA group). Voriconazole plasma levels will be measured on day 1 (both peak and trough levels), day 3, day 5, day 10, and day 14 (all trough levels). For CA group patients, voriconazole dosage will be adjusted according to the trough levels of day 5 (steady-state level). Predefined dose adjustment protocol will be used (< 1 µg/ml: 50% increase, 1~5.5 µg/ml: no change, > 5.5 µg/ml: 50% decrease). For EA group patients, voriconazole dosage will be adjusted according to the each measurements of voriconazole levels from day 1. Adjusted dosage will be calculated using the NONMEN software.

SUMMARY:
Voriconazole, a newer triazole-derivative, has become the drug of choice for many invasive fungal infections, including invasive Aspergillosis. Recently, therapeutic drug monitoring of voriconazole has been issued because of wide variations and unpredictability of voriconazole blood concentration. The objective of this study is 1) to characterize the pharmacokinetics of voriconazole in ICU patients on voriconazole prophylaxis or treatment, and 2) to develop and evaluate the prediction and adjustment models for voriconazole plasma levels.

DETAILED DESCRIPTION:
Patients will be randomly assigned into 2 groups: conventional adjustment group (CA group) and early adjustment group (EA group). Voriconazole plasma levels will be measured on day 1 (both peak and trough levels), day 3, day 5, day 10, and day 14 (all trough levels). For CA group patients, voriconazole dosage will be adjusted according to the trough levels of day 5 (steady-state level). Predefined dose adjustment protocol will be used (< 1 µg/ml: 50% increase, 1~5.5 µg/ml: no change, > 5.5 µg/ml: 50% decrease). For EA group patients, voriconazole dosage will be adjusted according to the each measurements of voriconazole levels from day 1. Adjusted dosage will be calculated using the NONMEN software. The target range of trough level is between 1.0 µg/ml and 5.5 µg/ml. The appropriateness of voriconazole level (day 5, day 10, and day 14), mortality, ICU stay, and the frequency of voriconazole-related adverse events will be compared. CYP2C19 polymorphism will be analyzed for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received voriconazole

Exclusion Criteria:

* Patients allergic to azole(s)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Appropriateness of voriconazole trough level | Day 3, day 5, day 10, and day 14

SECONDARY OUTCOMES:
Mortality | 2 week, 4 week, 8 week, 12 week, and 24 week
Voriconazole-related adverse event | 1 week, 2 week

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Ho Choi, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea